CLINICAL TRIAL: NCT02517658
Title: Adenotonsillectomy Postoperative Parental Teaching Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Khan (Other)
Responsible Party: Sponsor-Investigator, Sarah Khan, Clinical Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-00063
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-08

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Discharge Teaching (Active Comparator): Parents will receive standard discharge teaching from the nurse prior to discharge.
  Interventions: Other: Standard discharge teaching
- Video w/ post exam immediately after video (Experimental): Parents will watch the video and then take the post test immediately after watching the video.
  Interventions: Other: Video
- Video w/ post exam after discharge teaching (Experimental): Parents will watch the video but wait to take the post exam until after the discharge instructions are given by the nurse prior to discharge.
  Interventions: Other: Video; Other: Standard discharge teaching

INTERVENTIONS:
Other: Video — Watching a YouTube video containing post tonsillectomy discharge instructions.
  Arms: Video w/ post exam after discharge teaching; Video w/ post exam immediately after video
Other: Standard discharge teaching — Receiving standard post tonsillectomy discharge instructions from the nurse prior to discharge.
  Arms: Standard Discharge Teaching; Video w/ post exam after discharge teaching

SUMMARY:
The study will involve parents filling out a survey before & after watching a teaching tool video (https://www.youtube.com/watch?v=rIH63jqvlio) in addition to standard post-op teaching. The parents randomized to the video arms will watch the video while their child is in the OR and then either take the post survey immediately after or wait to take the survey until just prior to discharge. Parents not in the video arms of the study will also be asked to complete a survey pre and post standard pain management teaching.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregiver of any child having either adenotonsillectomy or tonsillectomy.

Exclusion Criteria:

* Non-english speaking families that require an interpreter.
* Any parent/family/caregiver that declines to be part of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Khan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Discharge Teaching | Video w/ Post Exam Immediately After Video | Video w/ Post Exam After Discharge Teaching
Started | 33 | 33 | 33
Completed | 33 | 33 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Discharge Teaching | Video w/ Post Exam Immediately After Video | Video w/ Post Exam After Discharge Teaching | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 33 | 33 | 99
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Female, Male data were not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Difference in Answers to Pre & Post Teaching Questionnaires
Description: Assessing the difference in how parents answered the questionnaire before receiving any discharge instructions and the questionnaire after watching the video or receiving standard discharge instructions by the nurse. Parents completed pre-instruction and post-instruction assessments of their knowledge of post-operative pain management, with responses scored on a 0-8 scale by assigning 1 point to each correct response out of 8 multiple-choice questions. Higher difference score means that the parents answered more questions correctly after the teaching/video.
Time Frame: approx. 1 - 2 hrs post-op
Measure: Median (Inter-Quartile Range); unit: difference in testing scores
Arm/Group | Standard Discharge Teaching | Video w/ Post Exam Immediately After Video | Video w/ Post Exam After Discharge Teaching
Number analyzed (Participants) | 33 | 33 | 33
difference in testing scores | -1 [-2 to 0] | 0 [-1 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: 72 hours post-op.
Arm/Group | Standard Discharge Teaching | Video w/ Post Exam Immediately After Video | Video w/ Post Exam After Discharge Teaching
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes